CLINICAL TRIAL: NCT04129398
Title: A Phase 3, Open-Label, Single-Arm Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of MK-8228 (Letermovir) for the Prevention of Human Cytomegalovirus (CMV) Infection and Disease in Adult Japanese Kidney Transplant Recipients
Brief Title: MK-8228 (Letermovir) in the Prevention of Human Cytomegalovirus (CMV) Infection and Disease in Adult Japanese Kidney Transplant Recipients (MK-8228-042)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8228-042; MK-8228-042 (Other: Merck Protocol Number); 195020 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus Infection; Cytomegalovirus Disease
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Letermovir (Experimental): Letermovir oral or intravenous (IV) formulation will be administered once daily for up to 28 weeks, beginning up to 7 days post-transplant. The dose will be 240 mg once daily for participants receiving concomitant cyclosporin A (CsA) and 480 mg once daily for participants not receiving CsA. IV infusion will be administered only to participants who are unable to swallow tablets or who have a condition that may interfere with absorption of the tablets.
  Interventions: Drug: Letermovir tablet; Drug: Letermovir IV

INTERVENTIONS:
Drug: Letermovir tablet — A single 240 mg tablet or two 240 mg tablets letermovir administered orally, once daily for 28 weeks
  Other Names: MK-8228; PREVYMIS®
Drug: Letermovir IV — IV solution of 240 mg (one vial) or 480 mg (2 vials) letermovir in 250 mL infused over 60 minutes, once daily for 28 weeks
  Other Names: MK-8228; PREVYMIS®

SUMMARY:
This study aims to evaluate the safety, efficacy and pharmacokinetics (PK) of Letermovir (LET) administered as prevention of cytomegalovirus (CMV) infection and disease in adult Japanese kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Meets recipient and/or donor CMV Immunoglobulin G (IgG) serostatus.
* Anticipates receiving a primary or secondary allograft kidney at the time of screening and have received a primary or secondary allograft kidney at the time of allocation.
* Is within 0 (i.e., day of transplantation) to 7 days (inclusive) post-kidney transplant at the time of allocation.
* Is a Japanese male or female from 18 years to any years of age inclusive, at the time of signing the informed consent.
* Female is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP); but if a WOCBP, she is using an acceptable contraceptive method, or is abstinent from heterosexual intercourse, and must have a negative highly sensitive pregnancy test within 72 hours before the first dose of study intervention.

Exclusion Criteria:

* Has received a previous solid organ transplant or hematopoietic stem cell transplant (HSCT).
* Is a multi-organ transplant recipient (e.g., kidney-pancreas).
* Has a history of CMV disease or suspected CMV disease within 6 months prior to allocation.
* Has positive results on CMV assay and/or CMV antigen test at any time between the completion of the transplant surgery and time of allocation.
* Has suspected or known hypersensitivity to active or inactive ingredients of LET formulations.
* Is on dialysis (for the purposes of this protocol dialysis includes hemofiltration) or plasmapheresis at the time of allocation.
* Has Child-Pugh Class C severe hepatic insufficiency at screening.
* Has post-transplant renal function of creatinine clearance (CrCl) ≤10 mL/min at allocation (measured locally).
* Has both moderate hepatic insufficiency AND moderate-to-severe renal insufficiency at screening.
* Has any uncontrolled infection on the day of allocation.
* Has documented positive results for human immunodeficiency virus antibody (HIV-Ab) test at any time prior to allocation, or for hepatitis C virus antibody (HCV-Ab) and with detectable HCV RNA within 90 days prior to allocation or hepatitis B surface antigen (HBsAg) within 90 days prior to allocation.
* Requires mechanical ventilation, or is hemodynamically unstable, at the time of allocation.
* Has a history of malignancy ≤5 years prior to signing informed consent.
* Has received within 30 days prior to allocation or plans to receive during the study any of the following: CMV immune globulin; any investigational CMV antiviral agent/biologic therapy.
* Has received any dose of LET prior to allocation.
* Has received within 7 days prior to allocation or plans to receive during the study any anti-CMV drug therapy.
* Is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Is taking or plans to take any of the prohibited medications listed in the protocol.
* Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5× half-life of the investigational compound.
* Has previously participated in this study or any other study involving LET.
* Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.
* Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 28 days following cessation of study therapy.
* Is expecting to donate eggs starting from the time of consent through at least 28 days following cessation of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- Japan (4):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital ( Site 0002), Nagoya, Aichi-ken
  - Sapporo City General Hospital ( Site 0004), Sapporo, Hokkaido
  - Osaka University Hospital ( Site 0003), Suita, Osaka
  - Tokyo Women's Medical University Hospital ( Site 0001), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ishida H, Goto N, Imamura R, Sasaki H, Unagami K, Futamura K, Murata Y, Oshima N, Eto T, Haber B. Letermovir safety and efficacy for cytomegalovirus prophylaxis in adult Japanese kidney transplant recipients: a multicenter, open-label, noncomparative Phase 3 study. Clin Exp Nephrol. 2024 Aug;28(8):822-831. doi: 10.1007/s10157-024-02471-0. Epub 2024 Apr 13. PMID 38615067
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult Japanese kidney transplant recipients who are organ donor (D) or organ recipient (R) seropositive (D+/R-, D+/R+ or D-/R+) for Cytomegalovirus (CMV) as participants.
Pre-assignment Details: Intravenous (IV) infusion of letermovir (LET) was intended to administer participants who cannot tolerate swallowing oral letermovir and/or does develop a condition that may interfere with the absorption of the oral LET. None of the participants received IV LET.
Groups:
- Letermovir: Letermovir oral or intravenous (IV) formulation was administered once daily for up to 28 weeks, beginning up to 7 days post-transplant. The dose was 240 mg once daily for participants receiving concomitant cyclosporin A (CsA) and 480 mg once daily for participants not receiving CsA. IV infusion was administered only to participants who were unable to swallow tablets or who had a condition that may have interfered with absorption of the tablets.
Period: Overall Study
Arm/Group | Letermovir
Started | 22
Completed | 20
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Letermovir
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with one or more adverse events (AEs)
Time Frame: Up to week 52 post-transplant
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 22
Percentage of Participants | 90.9

2. Primary Outcome: Percentage of Participants Who Discontinued From Study Drug Due to an AE
Description: Percentage of participants who discontinued from study drug due to an AE
Time Frame: Up to week 28 post-transplant
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir
Number analyzed (Participants) | 22
Percentage of participants | 13.6

3. Secondary Outcome: Percentage of Participants With Adjudicated CMV Disease or Undergone Anti-CMV Treatment
Description: CMV disease was defined as the presence of either CMV end-organ disease or CMV syndrome and was confirmed by an independent, blinded Clinical Adjudication Committee (CAC). Only CAC-confirmed ("adjudicated") cases were included in percentage of participants who met the endpoint. Investigator-assessed cases which were not confirmed by the CAC were not included. Participants who have undergone anti-CMV treatment was defined as initiation of approved anti-CMV agents based on at least one positive cell on CMV antigenemia and/or quantifiable CMV DNA PCR assay performed locally.
Time Frame: Up to Week 52 post-transplant
Population: All allocated participants who received at least one dose of study treatment, who were organ donor (D) or organ recipient (R) seropositive (D+/R-, D+/R+ or D-/R+) for Cytomegalovirus (CMV) and had no detectable CMV viral DNA (measured by central laboratory) on Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Letermovir D+/R-: Letermovir oral or intravenous (IV) formulation was administered once daily for up to 28 weeks, beginning up to 7 days post-transplant. The dose was 240 mg once daily for participants receiving concomitant cyclosporin A (CsA) and 480 mg once daily for participants not receiving CsA. IV infusion was administered only to participants who were unable to swallow tablets or who had a condition that may have interfered with absorption of the tablets. Letermovir D+/R- represents the D+/R- subgroup.
- Letermovir R+: Letermovir oral or intravenous (IV) formulation was administered once daily for up to 28 weeks, beginning up to 7 days post-transplant. The dose was 240 mg once daily for participants receiving concomitant cyclosporin A (CsA) and 480 mg once daily for participants not receiving CsA. IV infusion was administered only to participants who were unable to swallow tablets or who had a condition that may have interfered with absorption of the tablets. Letermovir R+ represents the R+ subgroup (D+/R+ or D-/R+)
Arm/Group | Letermovir | Letermovir D+/R- | Letermovir R+
Number analyzed (Participants) | 21 | 12 | 9
Percentage of Participants
  With CMV Disease or Started Anti-CMV Treatment Through Week 28 Post-Transplant | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 33.6]
  With CMV Disease or Started Anti-CMV Treatment Through Week 52 Post-Transplant | 19.0 [5.4 to 41.9] | 33.3 [9.9 to 65.1] | 0.0 [0.0 to 33.6]

4. Secondary Outcome: Percentage of Participants With Adjudicated CMV Disease
Description: CMV disease was defined as the presence of either CMV end-organ disease or CMV syndrome and was confirmed by an independent, blinded Clinical Adjudication Committee (CAC). Only CAC-confirmed ("adjudicated") cases were included in percentage of participants who met the endpoint. Investigator-assessed cases which were not confirmed by the CAC were not included.
Time Frame: Up to Week 52 post-transplant
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir | Letermovir D+/R- | Letermovir R+
Number analyzed (Participants) | 21 | 12 | 9
Percentage of Participants
  With CMV Disease Through Week 28 Post-Transplant | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 33.6]
  With CMV Disease Through Week 52 Post-Transplant | 9.5 [1.2 to 30.4] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 33.6]

5. Secondary Outcome: Percentage of Participants With Quantifiable CMV DNAemia
Description: Quantifiable CMV DNAemia (central) was defined as any case with a numeric value or >910,000,000 (not including reporting of PCR results as "detected, not quantifiable") using the Roche COBAS® AmpliPrep/COBAS TaqMan® (CAP/CTM) assay, which was performed by the central laboratory.
Time Frame: Up to Week 52 post-transplant
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Letermovir | Letermovir D+/R- | Letermovir R+
Number analyzed (Participants) | 21 | 12 | 9
Percentage of participants
  Quantifiable CMV DNAemia Through Week 28 Post-transplant | 4.8 [0.1 to 23.8] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 33.6]
  Quantifiable CMV DNAemia Through Week 52 Post-transplant | 23.8 [8.2 to 47.2] | 41.7 [15.2 to 72.3] | 0.0 [0.0 to 33.6]

6. Secondary Outcome: Area Under the Concentration-time Curve During a Dosing Interval (AUCtau) of Plasma Letermovir-oral Treatment
Description: AUCtau was defined as a measure of letermovir exposure that was calculated as the product of plasma drug concentration and time following an oral administration of letermovir.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment and had at least one measurable pharmacokinetic (PK) sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Letermovir
Number analyzed (Participants) | 21
ng*hr/mL | 156000 (47.3)

7. Secondary Outcome: Trough Concentration (Ctrough) of Plasma Letermovir - Oral Treatment
Description: Ctrough was defined as the minimum concentration of letermovir that occurred immediately following an oral administration of letermovir.
Time Frame: Any day between Days 6-10: 24hrs post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment and had at least one measurable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Letermovir
Number analyzed (Participants) | 21
ng/mL | 1700 (121.9)

8. Secondary Outcome: Maximum Concentration (Cmax) of Plasma Letermovir - Oral Treatment
Description: Cmax was defined as the maximum concentration of letermovir observed in plasma following an oral administration of letermovir.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Letermovir
Number analyzed (Participants) | 21
ng/mL | 17900 (31.1)

9. Secondary Outcome: Time to Reach Cmax (Tmax) of Plasma Letermovir - Oral Treatment
Description: Tmax was defined as the time required post dosing to reach a maximum plasma concentration of letermovir following an oral administration of letermovir.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | Letermovir
Number analyzed (Participants) | 21
hr | 2.50 [0.92 to 23.35]

10. Secondary Outcome: Apparent Clearance at Steady State (CLss/F) of Plasma Letermovir - Oral Treatment
Description: Apparent clearance at steady state (CLss/F) of plasma letermovir following an oral administration of letermovir.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Letermovir
Number analyzed (Participants) | 21
L/hr | 3.08 (47.3)

11. Secondary Outcome: Area Under the Concentration-time Curve During a Dosing Interval (AUCtau) of Plasma Letermovir - IV Treatment
Description: AUCtau was defined as a measure of letermovir exposure that was calculated as the product of plasma drug concentration and time following an IV administration of letermovir was intended to measure.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment and had at least one measurable PK sample. None of the participants received letermovir IV.
Arm/Group | Letermovir
Number analyzed (Participants) | 0

12. Secondary Outcome: Trough Concentration (Ctrough) of Plasma Letermovir - IV Treatment
Description: Ctrough was defined as the minimum concentration of letermovir that occurred immediately following an IV administration of letermovir was intended to measure.
Time Frame: Pre-dose on Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, 24 and 28
Population: as for outcome 11
Arm/Group | Letermovir
Number analyzed (Participants) | 0

13. Secondary Outcome: Concentration at the End of Infusion (Ceoi) of Plasma Letermovir - IV Treatment
Description: Ceoi is defined as the amount of letermovir in plasma following an IV administration of letermovir was intended to measure.
Time Frame: Any day between Days 6-10: at end of infusion (1 hours post dose)
Population: as for outcome 11
Arm/Group | Letermovir
Number analyzed (Participants) | 0

14. Secondary Outcome: Clearance at Steady State (CLss) of Plasma Letermovir - IV Treatment
Description: Clearance at steady state (CLss) of plasma letermovir following an IV administration of letermovir was intended to measure.
Time Frame: Any day between Days 6-10: pre-dose, 1, 2.5, 5, 8 and 24 hrs post-dose
Population: as for outcome 11
Arm/Group | Letermovir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to week 52 post-transplant
Description: All-Cause Mortality included all randomized participants. Non-serious and SAEs were reported for all randomized participants who received at least one dose of study treatment.
Arm/Group | Letermovir
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=22)
Constipation (Gastrointestinal disorders) | 1 (1)
Adenoviral haemorrhagic cystitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04129398/Prot_SAP_000.pdf